CLINICAL TRIAL: NCT02377050
Title: Randomized Controlled Trial of Higher-Volume Feedings in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Colm Travers, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UAB NEO 013
Record Dates: First submitted 2014-12-01; First posted 2015-03-03 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Infant Premature
Keywords: Nutritional support
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher Volume Feeding Goal (Active Comparator): Infants randomized to this group will have higher volume feeding goals of 180-200 ml/kg/day.
  Interventions: Other: Higher Volume Feeding Goal
- Usual Volume Feeding Goal (No Intervention): Infants randomized to this group will have feeding goals of 140-160 ml/kg/day.

INTERVENTIONS:
Other: Higher Volume Feeding Goal — feeding volume goal of 180-200 ml/kg/day
  Arms: Higher Volume Feeding Goal

SUMMARY:
The primary hypothesis is that preterm infants who are less than or equal to 32 weeks gestation and weigh 1001-2500 grams at birth will have an increase in weight gain with a feeding goal of 180-200 ml/kg/day more than the commonly used feeding goal of 140-160 ml/kg/day

DETAILED DESCRIPTION:
The proposed trial is designed to test the primary hypothesis that in preterm infants weighing 1001-2500 grams at birth and who are less than or equal to 32 weeks gestation, feeding goals of 180-200 ml/kg/day will increase weight gain (g/k/day) from time of enrollment to discharge home or 36 weeks post-menstrual age (PMA)(whichever comes first) more than the commonly used feeding goal volume of 140-160 ml/kg/day (usual feeding goal). This is a pilot study to determine the safety of increased volumes of feedings as opposed to fortification of feedings.

ELIGIBILITY:
Inclusion Criteria:

* Inborn or outborn infants born at a gestational age of 32 weeks or less; Birthweight 1001-2500; Feeding volume of at least 120 ml/kg/day; Enrolled prior to 28 days of age and prior to exceeding 32 weeks

Exclusion Criteria:

* Hemodynamically significant patent ductus arteriosis; History of necrotizing enterocolitis Bell Stage II or greater; Known gastrointestinal or neurologic malformations; Prior or planned enrollment into the NICHD MILK Trial; Terminal illness or decision to withhold or limit support

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2015-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Weight gain | baseline to average 12 weeks of age
  Average change in weight between baseline and 12 weeks

SECONDARY OUTCOMES:
Mid arm circumference | baseline to average 12 weeks of age
  average change in mid arm circumference between baseline and 12 weeks
Length | baseline to average 12 weeks of age
  average change in length between baseline and 12 weeks
Head circumference | baseline to average 12 weeks of age
  average change in head circumference between baseline and 12 weeks
Caloric intake | 36 weeks
  Average difference in weekly caloric intake between groups
Length of stay | 36 weeks or discharge
  Days from study entry to discharge home
Rates of infants less than 10th percentile for weight | 36 weeks or discharge
  Rates of infants less than 10th percentile for weight at study completion
Change in weight z score | 36 weeks or discharge
  Change in weight z score from study entry to completion
Change in length z score | 36 weeks or discharge
  Change in length z score from study entry to completion
Change in head circumference z score | 36 weeks or discharge
  Change in head circumference z score from study entry to completion

OTHER OUTCOMES:
Body fat composition | 36 weeks or discharge
  Percentage of body fat composition
Rates of necrotizing enterocolitis (Bell Stage ≥ 2) | 36 weeks or discharge
  Safety outcome: Rates of necrotizing enterocolitis (Bell Stage ≥ 2)
Rates of feeding intolerance | 36 weeks or discharge
  Safety outcome: Rates of feeding intolerance defined as withholding feeds for > 24 hours due to gastrointestinal cause after study entry
Rates of culture proven sepsis | 36 weeks or discharge
  Safety outcome: Rates of blood culture positive sepsis after study entry
Duration of respiratory support | 36 weeks or discharge
  Safety outcome: Duration of respiratory support (oxygen, continuous positive airway pressure/high flow nasal cannula/mechanical ventilation) after study entry
Rates of bronchopulmonary dysplasia | 36 weeks or discharge
  Safety outcome: Rates of bronchopulmonary dysplasia
Rates of moderate to large or symptomatic patent ductus arteriosus | 36 weeks or discharge
  Safety outcome: Rates of moderate to large or symptomatic patent ductus arteriosus after study entry
Rates of adverse safety outcomes combined | 36 weeks or discharge
  Safety outcome: Safety outcome: Rates of bronchopulmonary dysplasia, necrotizing enterocolitis ≥ stage 2, feeding intolerance, culture proven sepsis, patent ductus arteriosus after study entry

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham; Colm Travers, MD, Principal Investigator — University of Alabama at Birmingham; Ariel A Salas, MD — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Salas AA, Travers CP, Jerome ML, Chandler-Laney P, Carlo WA. Percent Body Fat Content Measured by Plethysmography in Infants Randomized to High- or Usual-Volume Feeding after Very Preterm Birth. J Pediatr. 2021 Mar;230:251-254.e3. doi: 10.1016/j.jpeds.2020.11.028. Epub 2020 Nov 25. PMID 33248115
- [Derived] Travers CP, Wang T, Salas AA, Schofield E, Dills M, Laney D, Yee A, Bhatia A, Winter L, Ambalavanan N, Carlo WA. Higher- or Usual-Volume Feedings in Infants Born Very Preterm: A Randomized Clinical Trial. J Pediatr. 2020 Sep;224:66-71.e1. doi: 10.1016/j.jpeds.2020.05.033. Epub 2020 May 25. PMID 32464224